CLINICAL TRIAL: NCT00152165
Title: A Biomechanical Assessment of the DYNESYS Stabilization System Using Radiostereometric Analysis
Brief Title: Use of Radiostereometric Analysis (RSA) Following Spinal Fusion Versus the DYNESYS Stabilization System
Status: Completed | Type: Observational
Sponsor: State University of New York - Upstate Medical University (Other)
Collaborators: Zimmer Biomet (Industry)
Other Study IDs: SUNY UMU IRB# 4895
Record Dates: First submitted 2005-09-08; First posted 2005-09-09 (Estimated); Last update posted 2008-12-02 (Estimated); Status verified 2008-12

CONDITIONS: Spinal Fusion; Orthopedic Procedures
Keywords: spinal motion; tantalum beads; DYNESYS Stabilization system; spinal fusion; Radiostereometric Analysis following spinal fusion; Radiostereometric Analysis following surgery with DYNESYS Stabilization System

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Procedure: Radiostereometric Analysis beads inserted during surgery

SUMMARY:
Twelve subjects will be sought for this study. Six subjects will receive the DYNESYS system and six subjects will receive a posterior lumbar interbody fusion (PLIF) with the Silhouette device. All subjects will already be participating in the DYNESYS multi-center study (under IRB #4884) and will have been randomized to either group. Five tantalum beads will be inserted into each vertebra associated with the DYNESYS or fusion surgery. Subjects will be followed in conjunction with the multi-center follow-up schedule and will have RSA exams at the following time points after surgery: 3, 6, 12, 18, and 24 months. Standing neutral, flexion, extension, and lateral bending films will be collected at each time point and the amount of motion in each direction of the "marked" vertebrae will be measured. The time points have been selected based on their clinical relevance for comparison against the standard of care, which is the fusion procedure. Depending on the initial tension of the annular fibers, it is possible the DYNESYS will exhibit more motion with time. The time points are important to track the potential changes.

DETAILED DESCRIPTION:
The amount of motion of the vertebrae following spinal surgery is important in determining the success of a procedure. Assessment of spinal motion has been, and continues to be, a difficult clinical problem. Errors of up to 10 degrees for simple measurements of flexion, extension, and side bending have been recorded using conventional radiographs. It has therefore been difficult to accurately measure changes in spinal motion using conventional radiographs.

Radiostereometric Analysis, or RSA, is an accurate in vivo measurement technique using two simultaneous radiographs for examining spinal motion. The measurement accuracy offered by this technique far exceeds the manual techniques currently used. In addition to improved accuracy, it provides more information on spinal motion in comparison to conventional radiographs. Utilization of the RSA technology at the IHP and the United States is in its infancy. The investigators have placed much effort over the past 1-2 years to put the necessary dedicated resources and personnel in place. This has been a collaborative effort between the Department of Orthopedic Surgery and the Imaging Core at IHP. Preliminary work on the accuracy, reliability, and surgical planning for use of RSA has been completed and presented at national conferences.

The purpose of this study is to assess the amount of motion in the lumbar spine in patients with a dynamic stabilization system, DYNESYS. Currently the DYNESYS is under investigation as part of a multi-center clinical trial (IRB # 4884). The DYNESYS system is designed to allow for some motion in the spine while providing the necessary stability to the spinal segment. The amount and degree of this motion is currently unknown. By using tantalum bead markers placed in the spine at the time of the surgery, RSA analysis can determine the amount of motion the DYNESYS system provides. Normal spinal motion of the lower spine is approximately 18 and 12 degrees for flexion/extension and lateral bending, respectively. Lumbar interbody fusion, which is the current standard surgical procedure, results in 5 degrees or less of spinal motion. Since the DYNESYS provides dynamic stabilization, it is estimated that there will be a 20% loss of motion with the DYNESYS in comparison to normal motion. Two questions will be examined in this study: 1) what is the amount of flexion/extension and lateral bending motion that occurs in the spine with a dynamic stabilization system in relation to a lumbar interbody fusion procedure? and 2) will the amount of motion change during the time frame of the study?

This study will involve 12 patients (6 with DYNESYS and 6 with posterior lumbar interbody fusion, PLIF) here at SUNY Upstate Medical University. Any subject who is part of the DYNESYS multi-center clinical trial (IRB # 4884) will be approached to participate in this RSA study. The subjects will already have been randomly assigned to the fusion group or the DYNESYS group. The RSA study is a single center, non-randomized design. All 12 subjects will have 10-15 tantalum markers placed in their spine at the time of their DYNESYS or fusion surgery. After surgery, subjects will have the special x-rays taken and the RSA analysis will be completed. Subjects will be seen at the following time points after surgery: 3, 6, 12, 18, and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing spinal fusion
* Patients undergoing spinal surgery with DYNESYS Stabilization System

Exclusion Criteria:

* Pregnant women

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12
Dates: Start 2003-11

CONTACTS AND LOCATIONS:
Overall Officials: Nathaniel Ordway, MS, PE, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- Institute for Human Performance, Syracuse, New York, United States